CLINICAL TRIAL: NCT01246999
Title: Evaluation of the Effect of Age and Prior Immunity on the Response to Live or Inactivated Seasonal (A/California/7/2009-like, A/Perth/16/2009-like, and B/Brisbane/60/2008-like (B/Victoria Lineage) Influenza Vaccines in Children
Brief Title: Effect of Age and Prior Immunity to Response to Seasonal Influenza Vaccines in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John Treanor, M.D., University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URMC10-005/Dartmouth 22164
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Influenza; A/California/7/2009-like (2009 H1N1); A/Perth/16/2009-like (H3N2); B/Brisbane/60/2008-like (B/Victoria lineage)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Live Attenuated Influenza vaccine (Active Comparator): LAIV 0.2 ml will be given intranasally followed by LAIV 0.2 mg given intranasally 28 days later
  Interventions: Biological: Live attenuated Influenza vaccine
- Trivalent Influenza Vaccine 2010-2011 (Active Comparator): TIV will be given in a dose of .25mg 2 years to 36 months of age or .5 ml ages 37 months to 8 years intramuscularly followed by a second dose of .25mg 2 years to 36 months of age or .5 ml ages 37 months to 9 years intramuscularly 28 days later
  Interventions: Biological: Trivalent Influenza Vaccine
- TIV followed by LAIV (Active Comparator): TIV will be given in a dose of .25mg 2 years to 36 months of age or .5 ml ages 37 months to 9 years intramuscularly followed by LAIV given in a dose of .2 ml intranasally 28 days later
  Interventions: Biological: TIV followed by LAIV
- LAIV followed by TIV (Active Comparator): LAIV will be given in a dose of .2 ml intranasally followed by a dose of TIV given in a dose of .25 ml 2 years to 36 months or .5 ml 37 months to 9 years intramuscularly 28 days later
  Interventions: Biological: LAIV followed by TIV

INTERVENTIONS:
Biological: Live attenuated Influenza vaccine — 0.2 mL dose delivered through nasal spray, 0.1 ml in each nostril, 2 doses separated by 28 days
  Other Names: FluMist
  Arms: Live Attenuated Influenza vaccine
Biological: Trivalent Influenza Vaccine — .25 mL given intramuscularly to children 24 to 36 months of age, 2 doses given 28 days apart, .5 mL given intramuscularly to children 37 months to 9 years of age, 2 doses given 28 day s apart.
  Other Names: Seasonal Influenza Vaccine
  Arms: Trivalent Influenza Vaccine 2010-2011
Biological: TIV followed by LAIV — TIV .25 mL given intramuscularly to children 24 to 36 months of age or .5 mL given intramuscularly to children 37 months to 9 years of age, followed by FluMist 0.2 mL delivered by nasal spray (.1 mL in each nostril)28 days later
  Other Names: Seasonal Influenza Vaccines
  Arms: TIV followed by LAIV
Biological: LAIV followed by TIV — LAIV .2 mL given through nasal spray (.1 mL in each nostril) Followed by TIV .25 mL given intramuscularly to children 24 to 25 months of age or .5 mL given intramuscularly to children 36 months to 9 years of age 28 days later
  Other Names: Seasonal Influenza Vaccines
  Arms: LAIV followed by TIV

SUMMARY:
A total of 88 children between 2 and 9 years of age will be randomized to receive a two dose schedule of either licensed live attenuated trivalent seasonal influenza vaccine (LAIV) or licensed inactivated seasonal influenza vaccine (TIV)or TIV followed by LAIV or LAIV followed by TIV separated by 28 days. Children with a laboratory documented history of prior H1N1 infection will be excluded.

DETAILED DESCRIPTION:
The study will be conducted as a randomized, prospective, open-label evaluation of the clinical tolerability, vaccine virus shedding, and serum and mucosal antibody response to vaccination with either live trivalent influenza vaccine (LAIV) or trivalent influenza vaccine (TIV) in healthy children between the ages of 2 and 9 years. Children will be screened for antibody to A/Brisbane/57/07 (H1N1) and A/California/07/09 (H1N1), A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008 before and at indicated times after the start of the study. They will not be randomized based on antibody levels. Children with prior documented infection with the 2009 pandemic H1N1 virus will be excluded. Vaccine will be administered on days 0 and 28.

Safety of vaccination will be assessed using symptoms collected by parents for 7 days after each dose of vaccine. Serum will be obtained prior to and on day 28 following each dose of vaccine and assessed for antibody by HAI, ELISA, and neutralization techniques. Nasal secretions will be obtained by nasal wick prior to and on day 28 after each dose and assessed for HA-specific IgA (immune globulin A) and IgG (immune globulin G)antibody by ELISA. Nasal swabs will be obtained on days 2, 4, and 7 after each dose of live vaccine and assessed for the presence and magnitude of vaccine virus shedding of the live attenuated vaccine by rtRT-PCR (real-time reverse transcriptase polymerase chain reaction)and TCID50 (50% tissue culture infectious doses)on MDCK(Madin Darby Canine Kidney) cells.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 and 9 years, inclusive.
* No prior history of laboratory documented infection with novel H1N1 virus
* The subject must be in good health, as determined by: vital signs (heart rate <140 bpm; blood pressure: systolic ≥ 90 mm Hg and ≤140 mm Hg; diastolic ≤ 90 mm Hg; oral temperature <100.0ºF (fahrenheit); medical history; and targeted physical examination, when necessary, based on medical history. Stable medical condition is defined as: no recent increase in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months.
* The subject/parents are able to understand and comply with the planned study procedures, including being available for all study visits.
* The subject/parents have provided informed consent prior to any study procedures. (An assent will be obtained for all children as required by the institutional IRB (Institutional Review Board.)

Exclusion Criteria:

* Subjects with a laboratory documented history of previous novel H1N1 infection.
* History of egg allergy or allergy to other components of vaccine.
* History of wheezing.
* The subject is immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy.
* The subject has an active neoplastic disease.
* The subject has long-term (greater than 2 weeks) use of oral or parenteral steroids, or high-dose inhaled steroids (>800 mg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* The subject received immunoglobulin or another blood product within the 3 months prior to enrollment in this study.
* The subject has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days (or 56 days for vaccine naïve recipients).
* The subject has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include chronic conditions recognized as risk factors for influenza complications or as contraindications for live vaccination, including chronic cardiac (exclusive of hypertension) or pulmonary conditions (including asthma), diabetes mellitus, or renal impairment.
* The subject has an acute illness or an oral temperature greater than 99.9 degreesF (37.7 degrees C) within 3 days prior to enrollment or vaccination. Subjects who had an acute illness that was treated symptoms resolved are eligible to enroll as long as treatment is completed and symptoms resolve > 3 days prior to enrollment.
* The subject is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study, or intends to donate blood during the study period.
* The subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* The subject has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* The subject has a previous history of Guillain-Barré syndrome within 6 weeks of receipt of influenza vaccination.
* The subject has any condition that the principal investigator (PI) believes may interfere with successful completion of the study.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Treanor, M.D., Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Vaccine Research Unit Room 3-5000, Rochester, New York

REFERENCES:
- [Background] Hancock K, Veguilla V, Lu X, Zhong W, Butler EN, Sun H, Liu F, Dong L, DeVos JR, Gargiullo PM, Brammer TL, Cox NJ, Tumpey TM, Katz JM. Cross-reactive antibody responses to the 2009 pandemic H1N1 influenza virus. N Engl J Med. 2009 Nov 12;361(20):1945-52. doi: 10.1056/NEJMoa0906453. Epub 2009 Sep 10. PMID 19745214
- [Background] Shinde V, Bridges CB, Uyeki TM, Shu B, Balish A, Xu X, Lindstrom S, Gubareva LV, Deyde V, Garten RJ, Harris M, Gerber S, Vagasky S, Smith F, Pascoe N, Martin K, Dufficy D, Ritger K, Conover C, Quinlisk P, Klimov A, Bresee JS, Finelli L. Triple-reassortant swine influenza A (H1) in humans in the United States, 2005-2009. N Engl J Med. 2009 Jun 18;360(25):2616-25. doi: 10.1056/NEJMoa0903812. Epub 2009 May 7. PMID 19423871
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216
- [Background] Belshe RB, Edwards KM, Vesikari T, Black SV, Walker RE, Hultquist M, Kemble G, Connor EM; CAIV-T Comparative Efficacy Study Group. Live attenuated versus inactivated influenza vaccine in infants and young children. N Engl J Med. 2007 Feb 15;356(7):685-96. doi: 10.1056/NEJMoa065368. PMID 17301299
- [Background] Maassab HF. Biologic and immunologic characteristics of cold-adapted influenza virus. J Immunol. 1969 Mar;102(3):728-32. No abstract available. PMID 5773321
- [Background] Chanock RM, Murphy BR. Use of temperature-sensitive and cold-adapted mutant viruses in immunoprophylaxis of acute respiratory tract disease. Rev Infect Dis. 1980 May-Jun;2(3):421-32. doi: 10.1093/clinids/2.3.421. PMID 6997969
- [Background] Boyce TG, Gruber WC, Coleman-Dockery SD, Sannella EC, Reed GW, Wolff M, Wright PF. Mucosal immune response to trivalent live attenuated intranasal influenza vaccine in children. Vaccine. 1999 Aug 20;18(1-2):82-8. doi: 10.1016/s0264-410x(99)00183-8. PMID 10501238
- [Background] Sasaki S, Jaimes MC, Holmes TH, Dekker CL, Mahmood K, Kemble GW, Arvin AM, Greenberg HB. Comparison of the influenza virus-specific effector and memory B-cell responses to immunization of children and adults with live attenuated or inactivated influenza virus vaccines. J Virol. 2007 Jan;81(1):215-28. doi: 10.1128/JVI.01957-06. Epub 2006 Oct 18. PMID 17050593
- [Background] Cox RJ, Brokstad KA, Zuckerman MA, Wood JM, Haaheim LR, Oxford JS. An early humoral immune response in peripheral blood following parenteral inactivated influenza vaccination. Vaccine. 1994 Aug;12(11):993-9. doi: 10.1016/0264-410x(94)90334-4. PMID 7975853
- [Background] He XS, Holmes TH, Zhang C, Mahmood K, Kemble GW, Lewis DB, Dekker CL, Greenberg HB, Arvin AM. Cellular immune responses in children and adults receiving inactivated or live attenuated influenza vaccines. J Virol. 2006 Dec;80(23):11756-66. doi: 10.1128/JVI.01460-06. Epub 2006 Sep 13. PMID 16971435
- [Derived] Ilyushina NA, Haynes BC, Hoen AG, Khalenkov AM, Housman ML, Brown EP, Ackerman ME, Treanor JJ, Luke CJ, Subbarao K, Wright PF. Live attenuated and inactivated influenza vaccines in children. J Infect Dis. 2015 Feb 1;211(3):352-60. doi: 10.1093/infdis/jiu458. Epub 2014 Aug 26. PMID 25165161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the first year participants were randomly assigned to receive LAIV twice, TIV twice, LAIV followed by TIV or TIV followed by LAIV. In the second year, randomization was confined to 2 groups: LAIV twice or TIV followed by LAIV. 8/34 participants were in the two arms not included in the analysis.
Groups:
- LAIV - LAIV: LAIV 0.2 ml will be given intranasally followed by LAIV 0.2 mg given intranasally 28 days later
  Trivalent Seasonal Live attenuated Influenza vaccine: 0.2 mL dose delivered through nasal spray, 0.1 ml in each nostril, 2 doses separated by 28 days
- TIV - LAIV: TIV will be given in a dose of .25mg 2 years to 36 months of age or .5 ml ages 37 months to 9 years intramuscularly followed by LAIV given in a dose of .2 ml intranasally 28 days later
  Seasonal Influenza Vaccine TIV/LAIV: TIV .25 mL given intramuscularly to children 24 to 36 months of age or .5 mL given intramuscularly to children 37 months to 9 years of age, followed by FluMist 0.2 mL delivered by nasal spray (.1 mL in each nostril)28 days later
- LAIV - TIV: LAIV will be given intranasally followed by TIV intramuscularly
- TIV - TIV: TIV will be given IM followed by TIV IM
Period: Overall Study
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Started | 11 | 4 | 2 | 17
Completed | 11 | 3 | 2 | 15
Not Completed | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were confined to the children enrolled in the second year only. In the second year randomization was confined to the two groups of greatest interest: 1) LAIV IN twice and 2) IIV IM followed by LAIV IN.
Groups:
- TIV - TIV: TIV will be given followed by TIV 28 days later
- LAIV - TIV: LAIV will be given followed by TIV 28 days later
- Total: Total of all reporting groups
Arm/Group | LAIV - LAIV | TIV - LAIV | TIV - TIV | LAIV - TIV | Total
Number analyzed (Participants) | 11 | 4 | 17 | 2 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 4 | 17 | 2 | 34
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 5 | 1 | 10 | 0 | 16
  Male | 6 | 3 | 7 | 2 | 18
Region of Enrollment [Number; unit: participants]
  United States | 11 | 4 | 17 | 2 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Shedding Vaccine Virus of Each Subtype by PCR
Description: Nasal washes were collected on days 2, 4 and 7 after vaccination. Nasal swab specimens were tested for the presence of vaccine viruses by quantitative viral culture in MDCK cells at 33º C and by real-time quantitative reverse-transcriptase polymerase chain reaction (qRT-PCR) amplification. The limit of detection of vaccine viruses was 10^0.6 tissue culture infectious doses (50%)/ml for virus culture and 10^0.4 tissue culture infectious doses (50%)/ml for qRT-PCR.
Time Frame: baseline to day 7
Population: Outcome for shedding of live vaccine in all participants who received a live vaccine
Measure: Number; unit: participants
Groups:
- Trivalent Seasonal Live Attenuated Influenza Vaccine: LAIV 0.2 ml will be given intranasally followed by LAIV 0.2 mg given intranasally 28 days later
  Trivalent Seasonal Live attenuated Influenza vaccine: 0.2 mL dose delivered through nasal spray, 0.1 ml in each nostril, 2 doses separated by 28 days
- Seasonal Influenza Vaccine (TIV-LAIV): TIV will be given in a dose of .25mg 2 years to 36 months of age or .5 ml ages 37 months to 9 years intramuscularly followed by LAIV given in a dose of .2 ml intranasally 28 days later
  Seasonal Influenza Vaccine TIV/LAIV: TIV .25 mL given intramuscularly to children 24 to 36 months of age or .5 mL given intramuscularly to children 37 months to 9 years of age, followed by FluMist 0.2 mL delivered by nasal spray (.1 mL in each nostril)28 days later
- All First Dose Live Vaccine: All subjects who received LAIV as a first dose
Arm/Group | Trivalent Seasonal Live Attenuated Influenza Vaccine | Seasonal Influenza Vaccine (TIV-LAIV) | All First Dose Live Vaccine
Number analyzed (Participants) | 11 | 15 | 13
participants
  shedding H1N1 | 1 | 6 | 9
  shedding H3N2 | 1 | 5 | 9
  shedding B | 1 | 10 | 10

2. Secondary Outcome: Mean Peak H1N1 Virus Titer, Dose 1
Description: After the first dose of vaccine, the virus titer from nasal secretions was measured in tissue culture on days 2, 4 and 7 and the highest titer from one of those three time points was reported.
Time Frame: days 2, 4 and 7
Measure: Log Mean (Standard Deviation); unit: log10 TCID(50)/ml
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Number analyzed (Participants) | 11 | 3 | 2 | 15
log10 TCID(50)/ml | 1.8 (1.7) | 0.0 (0.0) | 1.4 (1.9) | 0.0 (0000)

3. Secondary Outcome: Mean Peak H3N2 Virus Titer, Dose 1
Description: as for outcome 2
Time Frame: days 2, 4 and 7
Measure: Log Mean (Standard Deviation); unit: log10 TCID(50)/ml
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Number analyzed (Participants) | 11 | 3 | 2 | 15
log10 TCID(50)/ml | 0.9 (1.6) | 0 (0) | 0 (0) | 0 (0)

4. Secondary Outcome: Mean Peak Influenza B Virus Titer, Dose 1
Description: as for outcome 2
Time Frame: days 2, 4 and 7
Measure: Log Mean (Standard Deviation); unit: log10 TCID(50)/ml
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Number analyzed (Participants) | 11 | 3 | 2 | 15
log10 TCID(50)/ml | 1.6 (2.0) | 0 (0) | 2.1 (2.9) | 0 (0)

5. Secondary Outcome: Mean Peak H1N1 Virus Titer, Dose 2
Description: After the second dose of vaccine, the virus titer from nasal secretions was measured in tissue culture on days 2, 4 and 7 and the highest titer from one of those three time points was reported.
Time Frame: days 2, 4 and 7
Measure: Mean (Standard Deviation); unit: log10 TCID(50)/ml
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Number analyzed (Participants) | 11 | 3 | 2 | 15
log10 TCID(50)/ml | 0.3 (0.99) | 0 (0) | 0 (0) | 1 (1.8)

6. Secondary Outcome: Mean Peak H3N2 Virus Titer, Dose 2
Description: as for outcome 5
Time Frame: days 2, 4 and 7
Measure: Mean (Standard Deviation); unit: log10 TCID(50)/ml
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Number analyzed (Participants) | 11 | 3 | 2 | 15
log10 TCID(50)/ml | 0.3 (0.9) | 0 (0) | 0 (0) | 0.3 (1.2)

7. Secondary Outcome: Mean Peak Influenza B Virus Titer, Dose 2
Description: as for outcome 5
Time Frame: days 2, 4 and 7
Measure: Mean (Standard Deviation); unit: log10 TCID(50)/ml
Arm/Group | LAIV - LAIV | TIV - LAIV | LAIV - TIV | TIV - TIV
Number analyzed (Participants) | 11 | 3 | 2 | 15
log10 TCID(50)/ml | 0 (0) | 0 (0) | 0 (0) | 1.3 (2)

ADVERSE EVENTS:
Groups:
- LAIV-LAIV: LAIV 0.2 ml will be given intranasally followed by LAIV 0.2 mg given intranasally 28 days later
  Trivalent Seasonal Live attenuated Influenza vaccine: 0.2 mL dose delivered through nasal spray, 0.1 ml in each nostril, 2 doses separated by 28 days
- TIV-LAIV: TIV will be given in a dose of .25mg 2 years to 36 months of age or .5 ml ages 37 months to 9 years intramuscularly followed by LAIV given in a dose of .2 ml intranasally 28 days later
  Seasonal Influenza Vaccine TIV/LAIV: TIV .25 mL given intramuscularly to children 24 to 36 months of age or .5 mL given intramuscularly to children 37 months to 9 years of age, followed by FluMist 0.2 mL delivered by nasal spray (.1 mL in each nostril)28 days later
- LAIV-TIV: LAIV will be given intranasally followed by TIV intramuscularly
- TIV-TIV: TIV will be given IM followed by IV IM
Arm/Group | LAIV-LAIV | TIV-LAIV | LAIV-TIV | TIV-TIV
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/2 | 0/17
Other Adverse Events (participants affected / at risk) | 8/11 | 3/15 | 1/2 | 12/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAIV-LAIV (N=11) | TIV-LAIV (N=15) | LAIV-TIV (N=2) | TIV-TIV (N=17)
runny nose (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 3
fever (General disorders) | 0 | 1 | 0 | 2
fatigue (General disorders) | 3 | 0 | 1 | 0
body ache (General disorders) | 0 | 0 | 0 | 2
headache (Nervous system disorders) | 0 | 0 | 0 | 1
eye redness (Eye disorders) | 1 | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 5
nose bleed (General disorders) | 0 | 1 | 0 | 1
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
ear ache (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
sore throat (Infections and infestations) | 1 | 1 | 0 | 1
stuffy nose (Infections and infestations) | 6 | 2 | 1 | 4
pain at the injection site (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 8
tenderness at the injection site (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 8
swelling at the injection site (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
redness at the injection site (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No